# **Clinical Study Protocol**

# Anti-platelet Precision Medicine to Prevent Stroke Early Progression and Recurrence (PRECISE)

**Protocol Number PRECISE** 

**Protocol Version** 3.1

**Version Date** July 23, 2018

Asan Medical Center and 21 Other **Study Center** 

Institutions

Dong-Wha Kang, Dept. of Neurology, Asan **Study Coordinator** 

**Medical Center** 

#### Confidentiality Statement

This document contains confidential information that must not be disclosed to anyone other than the principal investigator, investigators, the IRB and national regulatory authorities without prior written consent of the sponsor, except to obtain informed written consent to participate in the study from those providing the information of what is intended to be observed in the study.

# **\* PROTOCOL SYNOPSIS**

| Study title | Anti-platelet Precision Medicine to Prevent Stroke Early Progression and Recurrence (PRECISE) |
|---|---|
| Study phase and design | Pragmatic, multi-center, non-interventional, non-random trial based on prospective observational study |
| Study center | Asan Medical Center and 21 other institutions |
| Study coordinator | Dong-Wha Kang of Department of Neurology, Asan Medical Center |
| Study sponsor | Dong-Wha Kang of Department of Neurology, Asan Medical Center |
| Study funder | Chong Kun Dang Holdings |
| Study objectives | Primary objectives: To predict the clinical prognosis according to the antiplatelet treatment regime (aspirin as first-line treatment or in combination with clopidogrel), develop an AI that will search for and retrieve similar cases to each patient, and assess benefits of the technology: 1) To establish a stroke clinical-imaging library (big data) and develop Deep Learning-based AI that understands the relationship between anti-platelet agents and prognosis (progression or recurrence). AI will present the probability of stroke progression or recurrence following each treatment regime. AI will also help physicians make treatment decisions by searching for and retrieving existing cases with similar clinical conditions to the patients concerned. 2) To prove AI's merit in predicting prognosis by applying it to different patient groups. Secondary objective: To analyze practical results of antiplatelet agents: The aspirin alone group and the clopidogrel plus aspirin group will be compared against each other directly to help find the link between early progression and recurrence of stroke. Although this is a non-randomized trial, different statistical methodologies, including propensity score matching (PSM) should address confidence issues. |
| Study subjects | Acute ischemic stroke patients: Transient ischemic attack with confirmed acute ischemic stroke by brain imaging |

| <ol> <li>Inclusion criteria</li> <li>Male and/or female subjects who are aged 19 or over.</li> <li>Patients with acute noncardiac stroke or transient ischemic attack within hours of the onset (in the case of a transient ischemic attack, presented)</li> </ol> | . 70 |
|---|---|
| | . 70 |
| hours of the onset (in the case of a transient ischemic attack, present | 1/2 |
| | e of |
| ischemic/ischemic lesion on DWI or PWI). | |
| 3) Patients whose informed consent document within 72 hours of onset | was |
| signed and submitted. | |
| 4) Patients who were treated with aspirin alone or aspirin plus clopide | grel |
| resinate following stroke. | |
| Exclusion criteria 1) Patients who need anticoagulants for cardiac ischemic stroke or of | ther |
| reasons. | |
| 2) Patients who suffered severe stroke (National Institutes of Health St | roke |
| Scale> 16). | |
| 3) Patients who received emergency remission therapies such as tPA | and |
| thrombolysis. | |
| 4) Patients with neurological deterioration prior to signing an informed with the control of the | itten |
| consent document. | |
| 5) Patients who have undergone patency procedures (surgery or | tent |
| insertion) in the cerebrovascular or carotid arteries following stroke or | are |
| expected to do so. | |
| 6) Patients who are scheduled to undergo major surgery. | |
| 7) Patients who developed stroke during procedure/surgery. | |
| 8) Patients with recent history (in the past three months) of cere | |
| hemorrhage. | |
| 9) Patients with active internal bleeding. | |
| 10) Patients with severe anemia (Hb <10 g / dL) or bleeding tendency (pla | telet |
| <100,000 / uL or PT-INR> 1.7). | |
| 11) When a patient's life expectancy is less than 6 months due to other systems | emic |
| disease. | |
| Number of target Aspirin alone Aspirin + Clapidogral Total No. of | |
| study subjects Study subjects Glopidogrel target subjects resinate group | |
| No. of subjects 1,000 1,000 2,000 | |
| 1) Study duration: Approximately 36 months from IRB approval (subjection) | t to |
| Study duration change depending on subject enrollment speed) | |
| 2) Study duration for each subject: 90 days (± 15 days) | |
| Chindred Doubt of administration (does | |
| Study drug and Study drug Route of administration/dose Aspirin (monotherapy or 75~100mg once per day, initial loading dose) | of |
| dose concomitant therapy) 300~500mg/d is allowed | , i |

| | Clopidogrel resinate 75mg once per day, initial loading dose of (Concomitant therapy) 300mg/d is allowed |
|---|---|
| Study description | This is a pragmatic, multi-center, non-interventional, non-randomized prospective observational study. |
| | ■ Study procedures This is a prospective study of patients with acute stroke or transient ischemic |
| | attack within 72 hours of symptom onset. It is to mainly observe the patients' |
| | prognosis following the prescription of clopidogrel resinate and aspirin, collect relevant data and create big data for stroke. Based on this data, an AI, using |
| | various advanced statistical methodologies and deep learning techniques will be |
| | developed, and offer information regarding stroke prognosis by extracting |
| | markers that are characteristic of the relationship between stroke and the study |
| | drug. |
| | These analyses and results will include information on which drug regimen will |
| | better prevent the progression or recurrence of stroke by considering individual |
| | patient conditions. This is a pragmatic trial based on the prescription and |
| | treatment processes of routine clinical practice. Thus, there is no major restriction |
| | and with only the minimum exclusion criteria in place, it does not hinder usual |
| | clinical practices. Therefore, selecting and changing a patient's antiplatelet |
| | agents should be a rational medical judgment made by the patient's attending |
| | physician. The study will proceed without any major change in the sequence of |
| | routine clinical examinations, prescriptions, treatments, observations, etc. |
| | Provided, the process of storing and analyzing relevant information will be added to each study procedure in accordance with study methodologies and conditions |
| | no other special efforts or limitations will be required. |
| | The other special efforts of limitations will be required. |
| | The data will be collected prospectively, and the Al will generate brain imaging |
| | data and prognostic indicators for 3-months after stroke has occurred. The |
| | performance of the AI will be verified with independent test sets. |
| Dropout criteria | Because the subjects will receive usual stroke care practice, there will be no |
| | subject withdrawal or dropout due to issues related to the study description and |
| | design. |
| | However, if a research subject withdraws his/her consent to participate in the |
| | study (informed consent to have his/her personal information utilized), |
| | participation of the research subject will be suspended, and the data concerned |

will not be used in the study.

## **Endpoints**

#### Primary study endpoints

Al will learn and predict the occurrence of the following outcome variables (up to 3 months after stroke onset) according to the antiplatelet regimen (aspirin alone, or aspirin plus clopidogrel). An independent investigator, without knowledge of individual patient treatment regimens, will evaluate the same outcome variables separately and compare the results with those predicted by the Al:

- 1) Neurological deterioration
- 2) New ischemic stroke
- 3) Symptomatic hemorrhagic transformation of an ischemic stroke
- 4) Symptomatic intracranial hemorrhage
- 5) Myocardial infarction
- 6) Coronary revascularization without myocardial infarction
- 7) Major hemorrhage other than intracranial hemorrhage (life threatening or non-life-threatening)
- 8) Minor hemorrhage other than intracranial hemorrhage
- 9) Ischemic vascular death
- 10) Hemorrhagic vascular death
- 11) Other serious adverse events

#### Secondary study endpoints

A direct comparison between the aspirin alone group and the aspirin and clopidogrel combination therapy group for the incidence of 11 outcome variables evaluated by an independent investigator at the primary endpoints will be conducted.

# Statistical Methodology

### General principle

All the enrolled study subjects whose results are confirmed will be subject to analysis, and they will be selected and classified according to the study methodologies and objectives prior to analysis. During the study period, data will be regularly checked and managed so that the number of datasets and their levels will be maintained appropriately.

#### **Analyses of endpoints**

## Analysis of primary endpoints

1) The stroke clinical and imaging library (big data), that includes all the

- clinical/imaging information related to clinical prognoses, will be established, and based on a deep learning algorithm, AI that has learned the relationship between antiplatelet agents and the following prognostic information will be developed.
- 2) A probability of prognosis according to each treatment option prior to using antiplatelet agents will be offered. This information will help physicians select an antiplatelet agent by searching for and retrieving similar cases that match each patient.
- 3) The stroke clinic and imaging library (big data) regarding the effect of antiplatelet agents that are being prescribed mainly to stroke patients in the clinical setting and the prognostic information of the patients concerned will be constructed. The relationship and prognostic features of antiplatelet agents in preventing early progression and recurrence of stroke will be extracted and analyzed from the "Big Data."
- 4) The development of AI using deep learning techniques will provide the basis for analysis of internal and external variables of stroke. This technique will change the model composition in line with the features and numbers extracted from the data. The depth and structure of the model will segment and materialize the characteristics of the target subjects and will be accompanied by the optimal design and verification processes of the model to simultaneously consider clinical/image information.
- 5) The research analysis using the trained AI that will be developed will need to have its results clearly verified as to their quality/accuracy. The delivered outcome will be used directly or indirectly by physicians, but the performance and reliability of the results that will be generated are of significant importance. Therefore, the AI will learn and have its performance assessed based on the data that will continue to accumulate throughout this study. However, because of the features of deep learning technology, training and verification, using the same data may cause major issues such as overfitting. Therefore, a new dataset will be created to evaluate the performance of the AI.

#### Analysis of secondary endpoints

1) The propensity score matching (PSM) technique will be used to select either the aspirin monotherapy, or the clopidogrel resinate and aspirin combination therapy group which have matched important clinical/imaging parameters that affect the prognosis of stroke.

Confidential Page 6 of 38

| 2) | Compare prescriptio | h treatment | group | to | determine | whic |
|----|---------------------|-------------|-------|----|-----------|------|
| | · · · · · · | | | | | |